CLINICAL TRIAL: NCT05555316
Title: Prospective Single Arm Phase II Study of TACE Combined With Lenvatinib and MWA After Down-stage in the Treatment of Locally Advanced Large Hepatocellular Carcinoma
Brief Title: TACE Combined With Lenvatinib and MWA in the Treatment of Locally Advanced Large Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Huang Jinhua, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TALEM
Record Dates: First submitted 2022-01-20; First posted 2022-09-26 (Actual); Last update posted 2022-09-26 (Actual); Status verified 2022-09

CONDITIONS: Liver Tumor
Keywords: Large hepatocellular carcinoma; Lenvatinib; TACE; Microwave ablation
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE combined with Lenvatinib (Experimental): Three days after the first TACE treatment, when the liver function was evaluated as grade A / B, Lenvatinib was taken orally, 8mg / day (body weight less than 60kg) or 12mg / day (body weight equal to or more than 60kg).
  Interventions: Drug: TACE combined with Lenvatinib

INTERVENTIONS:
Drug: TACE combined with Lenvatinib — Three days after the first TACE treatment, when the liver function was evaluated as grade A / B, Lenvatinib was taken orally, 8mg / day (body weight less than 60kg) or 12mg / day (body weight equal to or more than 60kg). Lenvatinib reduction standard: 8mg / day; 4mg / day; 4mg, the next day.
  Other Names: lenvima

SUMMARY:
To explore the objective effectiveness and safety of TACE combined with Lenvatinib in the treatment of advanced liver cancer. After successful down-stage, radical microwave ablation was further performed.

DETAILED DESCRIPTION:
The purpose of this study is to explore the objective effective rate of TACE combined with Lenvatinib in the treatment of locally advanced liver cancer, so as to provide a new idea for the radical microwave ablation treatment mode after the decline of locally advanced liver cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years with hepatocellular carcinoma have an expected survival of at least 3 months;
* Number of tumors ≤ 3;
* Large hepatocellular carcinoma with tumor diameter ≥ 7 cm;
* Patients without inferior vena cava tumor thrombus, portal vein tumor thrombus and cholangiocarcinoma thrombus;
* Although there is arteriovenous fistula or arterioportal fistula, it can be completely blocked;
* Child Pugh grade A or B of liver function; ECoG physical fitness score < 2;
* No bleeding tendency, normal coagulation function or coagulation dysfunction can be corrected after treatment;
* Leukocyte count ≥ 3.0 × 109/L；
* Hemoglobin ≥ 8.5g/dl;
* Platelet count ≥ 50 × 109/L；
* The international normalized ratio of prothrombin time (INR) ≤ 2.3 or prothrombin time (PT) does not exceed the upper limit of normal control for 3 seconds;
* Serum creatinine was less than 1.5 times of the upper limit of normal;
* Patients and / or family members agree to join the clinical trial and sign the informed consent form

Exclusion Criteria:

* Diffuse hepatocellular carcinoma;
* Portal vein tumor thrombus;
* Combined with tumor thrombus of hepatic vein and inferior vena cava;
* Patients with lymph node metastasis and extrahepatic distant metastasis;
* The liver function was classified as child Pugh C and could not be improved by liver protection treatment;
* Arteriovenous fistula or arterioportal fistula with ineffective intervention;
* Uncorrectable coagulation dysfunction and obvious hemogram abnormalities, with obvious bleeding tendency;
* Intractable massive ascites;
* ECoG physical fitness score > 2 points;
* Combined with active infection, especially bile duct inflammation;
* Serious heart, lung, kidney, brain and other important organ diseases;
* Note: see attached table 1 for child Pugh classification of liver function; See attached table 2 for ECoG physical fitness score

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2019-11-10 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Down stage rate | 4 months
  if the patient achieve any of these three criteria： ① the patient was downgraded from BCLC stage C to BCLC stage B (portal branch tumor thrombus was inactive, the focus was less than or equal to 7cm; or the focus did not invade the surrounding tissue after shrinking) or Milan standard (single tumor diameter was not more than 5cm or less than or equal to 3 tumors, and the maximum diameter was not more than 3cm, without vascular invasion). ② Liver function reaches child Pugh grade A or B; ③ The patient is in good health and can tolerate ablation.

SECONDARY OUTCOMES:
RFS | 3 years
  Recurrence free survival indicates the length of time after MWA for a cancer ends that the patient survives without any signs or symptoms of HCC
Objective response rate | 3 years
  Change of the tumor size according to the modified response evaluation criteria in solid tumors (mRECIST) [see attached table 3], the efficacy is defined as CR (complete remission), PR (partial remission), SD (stable) and PD (Progress)
Changes of liver and kidney function | 3 years
  Changes of liver and kidney function index from blood biochemistry compared to baseline
TACE frequency and ablation frequency | 3 years
  To access the times and frequency of TACE and ablation

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Huang, Ph.D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No